CLINICAL TRIAL: NCT02110641
Title: Lifestyle, Exercise and Nutrition (LEAN) Study 2
Brief Title: Lifestyle, Exercise and Nutrition Study 2 (LEAN 2)
Acronym: LEAN 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1012007780_1
Record Dates: First submitted 2014-04-07; First posted 2014-04-10 (Estimated); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer; Weight Loss
Keywords: Breast Cancer; Survivorship; Weight Loss
MeSH Terms: conditions — Breast Neoplasms; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- In-Person or Telephone-Based Counseling (Active Comparator): The exact same information, content, schedule, and 30 minute sessions will be provided to telephone-based participants as offered to participants who receive in-person counseling. Participants will be taught diet, exercise and behavior change strategies via the telephone (weekly calls for month 1, every other week for months 2-3, and monthly for months 4-6). All lessons and diet and physical activity logs will be mailed to them at the beginning of the program. Participants will record their daily diet and exercise in the logs.
  Interventions: Behavioral: Weight Loss Counseling
- Usual Care/Wait List (No Intervention): At 6-months the participants in the Wait List group may choose to participate in the 11 sessions either in-person or via telephone or a combination of the two modes of delivery. They will also be offered the opportunity to return to Yale at 12-months (immediately after the end of the 6-month counseling sessions) to have weight and DEXA measured.

INTERVENTIONS:
Behavioral: Weight Loss Counseling — The intervention will be based on the Diabetes Prevention Program weight loss program, which uses a combination of reduced caloric intake, increased physical activity, and behavior therapy. The content of the weight loss program will be similar for the in-person and telephone interventions, but the approach will vary (i.e., in-person vs. telephone counseling). The weight loss intervention will be conducted by a Registered Dietitian, who has training in exercise physiology and behavior modification.
  Arms: In-Person or Telephone-Based Counseling

SUMMARY:
The specific aims of this study are to determine the efficacy and cost-effectiveness of a weight loss program compared with usual care (control) treatment on 6-month changes in body weight, body fat, serum hormones, and breast tissue markers associated with prognosis in breast cancer survivors.

DETAILED DESCRIPTION:
We will conduct a two-armed study comparing a combination of an in-person and telephone weight loss program compared to usual care/wait list in 100 breast cancer survivors. Women will be randomized into one of the study arms using a random permuted block design. Research staff collecting body composition data, as well as reviewing forms and entering data, will be blinded to the participant's study group.

ELIGIBILITY:
Inclusion Criteria:

* American Joint Committee on Cancer (AJCC) Stages 0-IIIC Breast Cancer
* BMI >25 kg/m2
* Completed surgery, chemotherapy and radiation at least 2 months ago
* Physically able to exercise
* Agrees to be randomly assigned to either weight loss or control
* Gives informed consent to participate in all study activities
* Able to come for baseline and 6-month clinic visits
* Mentally competent

Exclusion Criteria:

* Patients with double mastectomy

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index (BMI) | 6 months
  BMI will be calculated using weight and height measurements (weight (kg)/height (m)^2 ). Weight and height will be measured by research staff blinded to the participant's randomization group at baseline and 6-months. Participants will be weighed in light indoor clothing, without shoes, rounding up to the nearest 0.1 kg; height will be measured in a standard manner, without shoes, using a stadiometer, rounding up to the nearest 0.1 cm. All measures will be performed and recorded twice in succession.
Change in body weight in kilograms (kg) | 6 months
  Participants will be weighed in light indoor clothing, without shoes, rounding up to the nearest 0.1 kg. All measures will be performed and recorded twice in succession.
Change in percent body fat | 6 months
  Dual Energy X-Ray Absorptiometry (DEXA) scans will be performed at baseline and 6-months. The DEXA measurements will be made with a Hologic scanner (Hologic 4500 with a "Discovery" upgrade, Hologic Inc, Waltham, Mass). A whole-body scan takes approximately 10 minutes to complete. We will measure percent body fat utilizing DEXA.
Change in breast tissue markers | 6 months
  We will collect a breast tissue biopsy from the unaffected breast at baseline and 6 months. Six slides will be made from each specimen for immunohistochemistry, as follows: Ki67 (MIB-1, DAKO), IGF1 receptor (1D5; DAKO), insulin receptor (mouse anti-human monoclonal B1445; LifeSpan BioSciences), Estrogen receptor (SP1, NeoMarker), Progesterone receptor (pgR636, DAKO) and HER-2 neu (SP3, NeoMarker). Ki67 will be scored quantitatively (% positive nuclei) using the Aperio system (Specialized Histopathology Laboratory). Estrogen and progesterone receptors will be scored following current ASCO/CAP guidelines (percent positive, intensity). Her2 will be scored according to current ASCO/CAP guidelines (intensity of membrane staining). All other markers will be scored on a semi-quantitative scale (0 to 3+).

SECONDARY OUTCOMES:
Change in fasting insulin | 6 months
  All the hormones to be measured (insulin, IGF-1, leptin, adiponectin and C-reactive protein) have been previously measured in our lab and published. We will use immunoassay techniques and kits from Diagnostic Products Corporation (DPC, Los Angeles, CA) to measure each hormone value. Each woman's baseline and follow-up samples will be used in the same batch, and an equal number of intervention and control samples will also be included in the same batch. Blind duplicates are also included in and between batches to estimate coefficient of variations.
Change in Leptin | 6 months
  All the hormones to be measured (insulin, IGF-1, leptin, adiponectin and C-reactive protein) have been previously measured in our lab and published. We will use immunoassay techniques and kits from Diagnostic Products Corporation (DPC, Los Angeles, CA) to measure each hormone value. Each woman's baseline and follow-up samples will be used in the same batch, and an equal number of intervention and control samples will also be included in the same batch. Blind duplicates are also included in and between batches to estimate coefficient of variations.
Change in C-reactive protein | 6 months
  All the hormones to be measured (insulin, IGF-1, leptin, adiponectin and C-reactive protein) have been previously measured in our lab and published. We will use immunoassay techniques and kits from Diagnostic Products Corporation (DPC, Los Angeles, CA) to measure each hormone value. Each woman's baseline and follow-up samples will be used in the same batch, and an equal number of intervention and control samples will also be included in the same batch. Blind duplicates are also included in and between batches to estimate coefficient of variations.
Skin Carotenoids Assessment | 6 months
  Assessment of skin carotenoids will be done using Resonance RAMAN Spectroscopy (RRS). Briefly, a small scanner which shines blue light is placed on the palm of the hand for 30 seconds. The palm is cleaned with an alcohol wipe prior to the scan, A RRS reading is available after a further 30 seconds. The procedure is repeated at the same body location. Skin color is self assessed by the participants at the baseline visit using samples that are used in plastic surgery to assess skin color. Melanin content (skin color) may have a small effect on RRS, but this effect is minimized by assessing skin carotenoids in the palm, which has a lower melanin content than other body sites.
Maintenance of Weight Loss | 12 months
  A mailed follow up will be conducted at 12-months post randomization. Questionnaires will be mailed to the participant with a pre-paid envelope for their return. Information about current weight will be collected using this method.
Changes in salivary cortisol | 6 months
  Women will be asked to collect 3 saliva samples (wake up, midday and bedtime) for 4 days following the baseline biopsy visit and 6 month follow up visit. Samples will be collected using Salivettes for cortisol. The cotton ball is removed from the Salivette, chewed for 1 minute and returned to the Salivette. Samples will be refrigerated in the container provided. Samples will be returned by mail in a specialized self-addressed pre-paid envelope when sample collection is complete.

OTHER OUTCOMES:
Change in Physical Activity | 6 months
  The 7-Day Daily Activity Log (7-Day DAL) will be the primary measure used to compare physical activity levels at baseline and 6-months among the three groups. All participants will complete the log for seven consecutive days, recording the amount of time spent in moderate- to vigorous-intensity recreational exercise. We will calculate their total minutes per week of exercise. Participants randomized to in-person and telephone counseling will also complete the 7-day DAL weekly.
Change in Dietary Intake | 6 months
  The endpoint measures of diet change will be mean, group level changes in daily caloric intake, based on a 120-item food frequency questionnaire (FFQ) which was developed for the Women's Health Initiative Study and has been validated against 4-Day Food Records and 24-hour Dietary Recalls. FFQs will be administered at baseline and 6-months.

CONTACTS AND LOCATIONS:
Overall Officials: Melinda L Irwin, PhD, MPH, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Nguyen T, Irwin ML, Dewan AT, Cartmel B, Harrigan M, Ferrucci LM, Sanft T, Li F, Lu L, Salinas YD. Examining the effect of obesity-associated gene variants on breast cancer survivors in a randomized weight loss intervention. Breast Cancer Res Treat. 2021 Jun;187(2):487-497. doi: 10.1007/s10549-021-06151-5. Epub 2021 Mar 6. PMID 33677781